CLINICAL TRIAL: NCT02463435
Title: Effect of Nutritional Intervention and Olive Oil in Severe Obesity: Randomized Controlled Trial
Brief Title: Effect of Nutritional Intervention and Olive Oil in Severe Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Collaborators: Fundação de Amparo a Pesquisa do Estado de Goias (FAPEG) (Unknown); Unidade de Pesquisa Clinica (UPC) do Hospital das Clínicas/UFG (Unknown); Grupo de Estudos em Obesidade Grave (GEOG) (Unknown)
Responsible Party: Principal Investigator, Ana Paula dos Santos Rodrigues, Master in Nutrition and Health, Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 747.792
Record Dates: First submitted 2015-05-29; First posted 2015-06-04 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Severe Obesity
Keywords: nutritional management; olive oil; weight loss; body composition; nutrigenomics; polymorphisms; cardiovascular risk; sarcopenia; inflammation; food intake; sedentary lifestyle; patient adherence; bone density
MeSH Terms: conditions — Obesity, Morbid; Weight Loss; Sarcopenia; Inflammation; Sedentary Behavior; Patient Compliance | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nutritional intervention (Active Comparator): Patients under only nutritional intervention for weight loss
  Interventions: Behavioral: Nutritional intervention
- Nutritional intervention plus olive oil (Experimental): Patients under conventional treatment (nutritional intervention) plus extra virgin olive oil supplementation
  Interventions: Other: Nutritional intervention plus olive oil
- Olive oil (Experimental): Patient under habitual food consumption plus extra virgin olive oil supplementation
  Interventions: Dietary Supplement: Olive oil

INTERVENTIONS:
Behavioral: Nutritional intervention — Conventional treatment (Nutritional intervention) consists of prescription of individualized food plan to reduce 5 to 10% of initial body weight, nutritional counseling for comorbidities and promoting healthy eating habits and physical activity.
  Arms: Nutritional intervention
Other: Nutritional intervention plus olive oil — Nutritional intervention consists of prescription of individualized food plan to reduce 5 to 10% of initial body weight, nutritional counseling for comorbidities and promoting healthy eating habits and physical activity. Additionally, dietary supplementation with extra virgin olive oil (52 mL daily) will be held, divided in four (4) sachets per day, two (2) at lunch and two (2) at dinner.
  Arms: Nutritional intervention plus olive oil
Dietary Supplement: Olive oil — Patients will be instructed to maintain habitual food consumption and consume 52 mL of extra virgin olive oil daily in four (4) sachets per day, two (2) at lunch and two (2) at dinner.
  Arms: Olive oil

SUMMARY:
Obesity is a worldwide epidemic with increasing prevalence, specially severe obesity (Body Mass Index (BMI) ≥ 35 kg/m2). It is a multifactorial disease that involves genetic and environmental factors that lead to increased mortality from cardiovascular disease, diabetes, cancer, among others and impairs life quality. Most research on severe obesity focuses on surgical alternatives and their results, thus this clinical trial aims to evaluate the effect of a non-pharmacological approach based on nutritional intervention and supplementation with a functional food, the olive oil. It will analyze the effectiveness of interventions on: weight loss, improvements on body composition and inflammatory profile (TNF-alfa, interleucins 1, 6 and 10, adiponectin), insulin resistance and serum lipids control, changing eating habits and physical activity practice, modification on bone mineral density and sarcopenia, and reduction of cardiovascular risk and other diseases. Also, it will be investigated the influence of polymorphisms (Pro12Ala of PPAR-γ gene, -174G>C of IL6 gene e Trp64Arg of ADRB3 gene) on nutritional intervention effectiveness with and without olive oil. This research looks for improving severely obese patient's care and contributing to effective results by reducing costs and risk treatment. The investigators believe that this informations will contribute significantly to the scientific field, expanding the knowledge about severe obesity.

DETAILED DESCRIPTION:
After enrollment, patients undergo a diagnostic phase (baseline) with nutritional, anthropometric and body composition assessment (multifrequency bioelectrical impedance analysis and dual X-ray absorptiometry); investigation of clinical history; collecting blood samples; carotid artery intima-media thickness, heart rate variability and accelerometry assessments; and application of validated questionnaires to evaluate secondary outcomes. Patients will be randomized into three different treatment groups. Randomization will be stratified according to Body Mass Index (BMI) (BMI between 35 and 39,99 kg/m2 and BMI ≥ 40 kg/m2), allocation ratio 1:1:1 and parallel intervention. Then, trained nutritionists will deliver the intervention according to the patient group and they will be followed-up for 12 weeks, with visits each 4 weeks.

Interventions will be provided as follow:

Olive oil group: in order to evaluate the effect of only the extra virgin olive oil on primary and secondary outcomes, patients will be instructed to maintain habitual food consumption and consume 52 mL of extra virgin olive oil daily (4 sachets per day, 2 at lunch and 2 at dinner).

Nutritional intervention group: patients assigned to this group will receive nutritional intervention consisting of prescription of individualized food plan to reduce 5 to 10% of initial body weight, nutritional counseling for comorbidities and promoting healthy eating habits and physical activity. Resting Energy Expenditure (REE) will be calculated according to Horie-Waitzberg & Gonzalez equation developed for severe obese individual using current weight and lean body mass (Horie et al., 2011). Total energy expenditure (TEE) will be calculated multiplying REE by activity factor recommended by Institute of Medicine (Trumbo et al., 2005) and thermic effect of food (Hill, Wyat, Peters, 2012). Total energy value (TEV) of diet will be determined reducing 550 to 1100 kcal from TEE to reach 0.5 to 1.0 weekly weight reduction according to the patient's individual goal. Distribution of macronutrients will follow Dietary Reference Intake (DRI) recommendation: 45-65% of carbohydrates, 10-35% of proteins and 20-35% of lipids (Trumbo et al., 2002). Fat acids (FA) will be distributed as recommended by Sociedade Brasileira de Cardiologia (Sposito et al., 2007): ≤ 7% saturated FA, ≤ 20% monounsaturated FA and ≤ 7% polyunsaturated FA. Food plan prescription will distribute TEV in 4-6 meals. Motivation will be held to changing eating and lifestyle habits.

Nutritional intervention plus olive oil: this group will receive conventional intervention plus supplementation of 52 mL of extra virgin olive oil daily (4 sachets per day, 2 at lunch and 2 at dinner).

At the end of follow-up the same assessments performed at diagnostic phase will be held.

To detect a reduction of 10 kg, with standard deviation of 30, which is in agreement with the study of Rodrigues e Silveira (2011), with a two-sided 5% significance level and a power of 80%, a sample size of 50 patients per group will be necessary, given an anticipated dropout rate of 42,9%.

This research will be conducted at a capital of center Brazil, at Unidade de Pesquisa Clínica of Hospital das Clínica/UFG, Faculty of Medicine/UFG.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥ 35 kg/m2
* Residence in Goiânia or metropolitan area
* Patients referred by Secretaria Municipal de Saúde to Severe Obese Nutrition Clinic

Exclusion Criteria:

* To have already performed bariatric surgery
* Pregnancy
* Reduction greater than 8% of body weight in the past 3 months
* To have been treated at Severe Obesity Nutrition Clinic or have received nutritional counseling in another place in the last 2 years
* Anti-obesity drugs use
* Regular utilization of anti-inflammatory drugs or corticosteroids
* HIV/AIDS, heart failure, kidney failure, hepatic insufficiency, chronic obstructive pulmonary disease and cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2015-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Anthropometric measurements change | Baseline, week 12
  Measurements of weight, arm circumference and Body Mass Index (BMI) will be evaluated to assess anthropometric change.
Body composition change | Baseline, week 12
  Body fat mass (BFM), body fat percentage (%BF) and body mass density (BMD) will be evaluated to assess body composition change. BFM and %BF will be assessed using multifrequency bioelectrical impedance analysis (BIA) and dual energy X-ray absorptiometry (DXA) and BMD will be assessed using DXA.

SECONDARY OUTCOMES:
Change in inflammation parameters | Baseline, week 12
  TNF-alfa
Change in inflammation parameters | Baseline, week 12
  Interleucin 6 (IL6), IL1, IL10
Change in inflammation parameters | Baseline, week 12
  Adiponectin
Change in inflammation parameters | Baseline, week 12
  C-reactive protein (CRP)
Change in inflammation parameters | Baseline, week 12
  Neutrophil to lymphocyte ratio (NLR) and lymphocyte to monocyte ratio (LMR)
Change in metabolic parameters | Baseline, week 12
  Lipid profile (total cholesterol, LDL-c, HDL-c, VLDL-c), insulin resistance (HOMA-IR, glycated hemoglobin), fasting glycaemia, hemogram
Change in kidney function | Baseline, week 12
  Creatinine, urea and uric acid
Change in liver function | Baseline, week 12
  AST and ALT
Change in thyroid function | Baseline, week 12
  TSH, T4 and parathyroid hormone
Change in vitamins | Baseline, week 12
  Vitamin D, vitamin B12 and folic acid
Change in minerals | Baseline, week 12
  Iron, calcium, sodium, potassium and zinc
Change in cardiovascular risk using Global Risk Score (GRS) | Baseline, week 12
Change in cardiovascular risk using Framingham Risk Score (FRS) | Baseline, week 12
Change in cardiovascular risk using heart rate variability (HRV) | Baseline, week 12
Change in cardiovascular risk using Homocystein level | Baseline, week 12
Polymorphism Pro12Ala of Peroxisome Proliferator-Activated Receptor Alfa (PPAR-alfa) | Baseline, week12
  Difference in responses between intervention groups for anthropometric measurements (weight, arm circumference and body mass index) and body composition variables (body fat mass and body fat percentage) according to this polymorphism
PolymorphismTrp64Arg of Beta-3 Adrenergic Receptor (ADRB3) gene | Baseline, week12
  Difference in responses between intervention groups for anthropometric measurements (weight, arm circumference and body mass index) and body composition variables (body fat mass and body fat percentage) according to this polymorphism
Polymorphism -174G>C of Interleukin 6 (IL6) gene. | Baseline, week12
  Difference in responses between intervention groups for anthropometric measurements (weight, arm circumference and body mass index) and body composition variables (body fat mass and body fat percentage) according to this polymorphism
Change in physical activity practice using Global Physical Activity Questionnaire | Baseline, week 12
Change in physical activity practice using accelerometry | Baseline, week 12
Change in food intake using Food Frequency Questionnaire | Baseline, week 12
Change in food intake using 24 hour recall | Baseline, week 12
Change in bone health parameters | Baseline, week 12
  Change in the following variables: bone density using DXA, falls and fractures and sun exposure
Change in obesity sarcopenia using muscle mass (evaluated using DXA) | Baseline, week 12
Change in obesity sarcopenia using handgrip strength | Baseline, week 12
Change in sarcopenia using usual gait speed | Baseline, week 12
Adherence to nutritional intervention | Baseline, week 12
  It will be evaluated through changes in food consumption (food frequency questionnaire)
Adherence to the health service | Baseline, week 12
  It will be evaluated through attendance to the clinic visits
Change in symptoms of anxiety and depression using Hospital Anxiety and Depression Scale | Baseline, week 12
Change in symptoms of binge eating disorderusing Binge Eating Disorder Scale | Baseline, week 12
Change in musculoskeletal pain using Visual Analog Scale | Baseline, week 12
Change in musculoskeletal pain using Nordic Musculoskeletal Questionnaire | Baseline, week 12

CONTACTS AND LOCATIONS:
Overall Officials: Erika A Silveira, PhD, Study Director — Universidade Federal de Goias - Faculdade de Medicina; Ana Paula S Rodrigues, MsC, Principal Investigator — Universidade Federal de Goias - Faculdade de Medicina; Jacqueline D Souza, MsC, Principal Investigator — Universidade Federal de Goias - Faculdade de Medicina; Camila KS Cardoso, MsC, Principal Investigator — Universidade Federal de Goias - Faculdade de Medicina; Lorena PS Rosa, MsC, Principal Investigator — Universidade Federal de Goias - Faculdade de Medicina; Annelisa SA Santos, MsC, Principal Investigator — Universidade Federal de Goias - Faculdade de Medicina; Andrea BS Canheta, MsC, Principal Investigator — Universidade Federal de Goias - Faculdade de Medicina; Carolina R Mendonça, MsC, Principal Investigator — Universidade Federal de Goias - Faculdade de Medicina
Locations (1):
- Unidade de Pesquisa Clínica do Hospital das Clínicas/UFG, Goiânia, Goiás, Brazil

REFERENCES:
- [Background] Hill JO, Wyatt HR, Peters JC. Energy balance and obesity. Circulation. 2012 Jul 3;126(1):126-32. doi: 10.1161/CIRCULATIONAHA.111.087213. PMID 22753534
- [Background] Horie LM, Gonzalez MC, Torrinhas RS, Cecconello I, Waitzberg DL. New specific equation to estimate resting energy expenditure in severely obese patients. Obesity (Silver Spring). 2011 May;19(5):1090-4. doi: 10.1038/oby.2010.326. Epub 2011 Jan 13. PMID 21233808
- [Background] Sposito AC, Caramelli B, Fonseca FA, Bertolami MC, Afiune Neto A, Souza AD, Lottenberg AM, Chacra AP, Faludi AA, Loures-Vale AA, Carvalho AC, Duncan B, Gelonese B, Polanczyk C, Rodrigues Sobrinho CR, Scherr C, Karla C, Armaganijan D, Moriguchi E, Saraiva F, Pichetti G, Xavier HT, Chaves H, Borges JL, Diament J, Guimaraes JI, Nicolau JC, dos Santos JE, de Lima JJ, Vieira JL, Novazzi JP, Faria Neto JR, Torres KP, Pinto Lde A, Bricarello L, Bodanese LC, Introcaso L, Malachias MV, Izar MC, Magalhaes ME, Schmidt MI, Scartezini M, Nobre M, Foppa M, Forti NA, Berwanger O, Gebara OC, Coelho OR, Maranhao RC, dos Santos Filho RD, Costa RP, Barreto S, Kaiser S, Ihara S, Carvalho Td, Martinez TL, Relvas WG, Salgado W; Sociedade Brasileira de Cardiologia. [IV Brazilian Guideline for Dyslipidemia and Atherosclerosis prevention: Department of Atherosclerosis of Brazilian Society of Cardiology]. Arq Bras Cardiol. 2007 Apr;88 Suppl 1:2-19. doi: 10.1590/s0066-782x2007000700002. No abstract available. Portuguese. PMID 17515982
- [Background] Trumbo P, Schlicker S, Yates AA, Poos M; Food and Nutrition Board of the Institute of Medicine, The National Academies. Dietary reference intakes for energy, carbohydrate, fiber, fat, fatty acids, cholesterol, protein and amino acids. J Am Diet Assoc. 2002 Nov;102(11):1621-30. doi: 10.1016/s0002-8223(02)90346-9. No abstract available. PMID 12449285
- [Derived] Rodrigues APDS, Batista SRR, Santos ASEA, Canheta ABS, Nunes BP, de Oliveira Rezende AT, de Oliveira C, Silveira EA. Multimorbidity and complex multimorbidity in Brazilians with severe obesity. Sci Rep. 2023 Oct 3;13(1):16629. doi: 10.1038/s41598-023-43545-5. PMID 37789121
- [Derived] Silveira EA, Rosa LPS, de Resende DP, Rodrigues APDS, da Costa AC, Rezende ATO, Noll M, de Oliveira C, Junqueira-Kipnis AP. Positive Effects of Extra-Virgin Olive Oil Supplementation and DietBra on Inflammation and Glycemic Profiles in Adults With Type 2 Diabetes and Class II/III Obesity: A Randomized Clinical Trial. Front Endocrinol (Lausanne). 2022 May 2;13:841971. doi: 10.3389/fendo.2022.841971. eCollection 2022. PMID 35586621
- [Derived] Longhi R, Santos ASEAC, Lopez-Yerena A, Rodrigues APS, Oliveira C, Silveira EA. The Effectiveness of Extra Virgin Olive Oil and the Traditional Brazilian Diet in Reducing the Inflammatory Profile of Individuals with Severe Obesity: A Randomized Clinical Trial. Nutrients. 2021 Nov 19;13(11):4139. doi: 10.3390/nu13114139. PMID 34836393
- [Derived] Kellen de Souza Cardoso C, Gondim Peixoto MDR, Dos Santos Rodrigues AP, Rodrigues Mendonca C, de Oliveira C, Aparecida Silveira E. Bone Mineral Density in Severely Obese Women: Health Risk and Health Protective Risk Factors in Three Different Bone Sites. Int J Environ Res Public Health. 2020 Sep 25;17(19):7017. doi: 10.3390/ijerph17197017. PMID 32992832
- [Derived] Canheta ABS, Santos ASEAC, Souza JD, Silveira EA. Traditional Brazilian diet and extra virgin olive oil reduce symptoms of anxiety and depression in individuals with severe obesity: Randomized clinical trial. Clin Nutr. 2021 Feb;40(2):404-411. doi: 10.1016/j.clnu.2020.05.046. Epub 2020 Jun 10. PMID 32675019
- [Derived] Aparecida Silveira E, Danesio de Souza J, Dos Santos Rodrigues AP, Lima RM, de Souza Cardoso CK, de Oliveira C. Effects of Extra Virgin Olive Oil (EVOO) and the Traditional Brazilian Diet on Sarcopenia in Severe Obesity: A Randomized Clinical Trial. Nutrients. 2020 May 21;12(5):1498. doi: 10.3390/nu12051498. PMID 32455620
- [Derived] Cardoso CKS, Santos ASEAC, Rosa LPS, Mendonca CR, Vitorino PVO, Peixoto MDRG, Silveira EA. Effect of Extra Virgin Olive Oil and Traditional Brazilian Diet on the Bone Health Parameters of Severely Obese Adults: A Randomized Controlled Trial. Nutrients. 2020 Feb 4;12(2):403. doi: 10.3390/nu12020403. PMID 32032997
- [Derived] Rodrigues APS, Rosa LPS, Silveira EA. PPARG2 Pro12Ala polymorphism influences body composition changes in severely obese patients consuming extra virgin olive oil: a randomized clinical trial. Nutr Metab (Lond). 2018 Jul 17;15:52. doi: 10.1186/s12986-018-0289-4. eCollection 2018. PMID 30026785